CLINICAL TRIAL: NCT03145389
Title: Effect of Continuous Thoracic Epidural Analgesia on Gut Motility Following Emergency Laparotomy for Intestinal Perforation Under General Anesthesia
Brief Title: Effect of Continuous Thoracic Epidural Analgesia on Gut Motility Following Emergency Laparotomy
Status: Completed | Type: Observational
Sponsor: Banaras Hindu University (Other)
Responsible Party: Principal Investigator, Dr Lal Dhar Mishra, Senior professor, Ex head of the department, Principal investigator, Department of Anesthesiology, Banaras Hindu University
Other Study IDs: EC/1683
Record Dates: First submitted 2017-04-25; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Analgesia, Epidural
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With epidural catheter placement: In this group of patients, after explaining about the procedure an 18 Gauge epidural catheter was placed in thoracic 11-12 inter vertebral space under strict asepsis.
  Interventions: Procedure: Epidural catheter placement
- Without epidural catheter placement: In this group of patients epidural catheter was not inserted and post operative pain was managed by using intravenous drugs.

INTERVENTIONS:
Procedure: Epidural catheter placement — After explaining about the procedure an 18 Gauge epidural catheter was inserted into thoracic 11-12 inter vertebral space under strict asepsis. Before inserting the epidural needle same space was infiltrated with adequate amount of 2% Lignocaine with Adrenaline (1: 200,000) to make the procedure pain free. Epidural space was confirmed by loss of resistance technique.
  Groups: With epidural catheter placement

SUMMARY:
Continuous thoracic epidural analgesia plays a very vital role in patients undergoing exploratory laparotomy. It not only supports a stable perioperative hemodynamics but also helps in early return of bowel activity.

DETAILED DESCRIPTION:
Intestinal perforation is one of the commonest surgical emergency that the investigators encounter in emergency. Perioperative management of most of such patients is a challenging task for the anesthesiologist, as patients are often hemodynamically unstable at the time of their presentation to emergency. Usual plan of anesthesia for these patients is general anesthesia with or without an epidural block. In routine practice the investigators often place an epidural catheter, primarily for postoperative analgesia, unless there is some contraindication to epidural analgesia. Most often lower thoracic epidural is preferred because of longer length of the laparotomy incision. Thoracic epidural analgesia with local anesthetic (LA) is not only effective in managing the post-operative pain; it is also helpful in supplementing intra-operative analgesia with reduced requirement of anesthetic, muscle relaxant and the analgesic (opioid) drugs. In addition, it has also been reported to be associated with early return of gut motility.

It appears that absent / significantly reduced pain leads to lesser stress response, leading to less sympathetic activation and lesser catecholamine release. As catecholamines are inhibitory to gastrointestinal motility, earlier return of gastro intestinal (GI) motility can be achieved by reducing perioperative pain by continuous epidural analgesia. Moreover, an effective epidural analgesia with LA results in avoidance of opioid analgesics for optimal perioperative pain relief, which too may be helpful in achieving earlier return of gut motility.

Thus the investigators aimed at determining the effect of continuous thoracic epidural analgesia on return of gut motility in patients undergoing emergency exploratory laparotomy following intestinal perforation and compare it with those in whom epidural analgesia was not used.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age 20-60 years
* Intestinal perforation posted for emergency exploratory laparotomy

Exclusion Criteria:

* Patient's refusal and uncooperativeness for epidural analgesia
* Hemodynamically unstable patients
* Patients with coagulation disorder
* Infection at the site of epidural insertion
* Spine deformity or spinal cord disease
* Raised intracranial pressure
* History of drug abuse
* Other comorbid conditions like diabetes mellitus, hypertension, thyroid disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Selected patients were randomly divided into two groups of 30 patients each,
  * Group-Ι : Epidural group
  * Group-ΙΙ: Non epidural group
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-03-20 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Return of bowel sound | Until 10th day after completion of surgery
  Earlier return of bowel sounds in epidural group

SECONDARY OUTCOMES:
Passage of flatus | Until 10th day after completion of surgery
  Earlier passage of flatus in epidural group
Feed tolerance | Until 10th day after completion of surgery
  Earlier feed tolerance in epidural group
Hospital discharge | Until 10th day after completion of surgery
  Earlier discharge from hospital in epidural group
Post operative pain | Until 10th day after completion of surgery
  Lesser pain in epidural group

CONTACTS AND LOCATIONS:
Overall Officials: Lal D Mishra, MD, PhD, Principal Investigator — Institute of Medical Sciences, Banaras Hindu University

IPD SHARING:
Plan to Share IPD: Undecided